CLINICAL TRIAL: NCT00806026
Title: Randomized, Double Blind, 12-Month Study Of Pregabalin In Subjects With Restless Legs Syndrome
Brief Title: Long Term Study Of Pregabalin In Idiopathic Restless Legs Syndrome Patients
Acronym: RLS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081186
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Results first posted 2012-09-27 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2012-08

CONDITIONS: Idiopathic Restless Legs Syndrome
Keywords: RLS
MeSH Terms: interventions — Pregabalin; Pramipexole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- PBO/PGB 300 mg (Experimental)
  Interventions: Drug: placebo and pregabalin
- PBO/PPX 0.25 mg (Active Comparator)
  Interventions: Drug: pramipexol
- PBO/PPX 0.5 mg (Active Comparator)
  Interventions: Drug: pramipexol
- PGB 300 mg (Experimental)
  Interventions: Drug: Pregabalin
- PPX 0.25 mg (Active Comparator)
  Interventions: Drug: pramipexol
- PPX 0.5 mg (Active Comparator)
  Interventions: Drug: pramipexol

INTERVENTIONS:
Drug: placebo and pregabalin — following 3 months placebo treatment, subjects are to be re-distributed to pregabalin 300 mg per day for 9 months. Both placebo and pregabalin are to be administered orally once a day, 1-3 hours before bedtime.
  Other Names: Lyrica
  Arms: PBO/PGB 300 mg
Drug: pramipexol — following 3 months placebo treatment, subjects are to be re-distributed to pramipexol 0.25mg per day for 9 months. Both placebo and pramipexol are to be administered orally once a day, 1-3 hours before bedtime.
  Other Names: Mirapex
  Arms: PBO/PPX 0.25 mg
Drug: pramipexol — following 3 months placebo treatment, subjects are to be re-distributed to pramipexol 0.5mg per day for 9 months. Both placebo and pramipexol are to be administered orally once a day, 1-3 hours before bedtime.
  Other Names: Mirapex
  Arms: PBO/PPX 0.5 mg
Drug: Pregabalin — pregabalin 300 mg, orally administered once a day, 1- 3 hours before the bedtime for 12 months
  Other Names: Lyrica
  Arms: PGB 300 mg
Drug: pramipexol — pramipexol 0.25 mg, orally administered once a day, 1- 3 hours before the bedtime for 12 months
  Other Names: Mirapex
  Arms: PPX 0.25 mg
Drug: pramipexol — pramipexol 0.5 mg, orally administered once a day, 1- 3 hours before the bedtime for 12 months
  Other Names: Mirapex
  Arms: PPX 0.5 mg

SUMMARY:
This purpose of this study is to investigate the efficacy and tolerability of pregabalin in treating idiopathic RLS patients for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic RLS with the presence of all four clinical manifestations of RLS
* RLS symptoms occur predominantly in the evening
* RLS history at least 6 months
* IRLS => 15 at the beginning and the end of placebo run-in
* Have =>15 nights with RLS symptoms in the month prior to screening

Exclusion Criteria:

* Any secondary RLS
* Current augmentation due to RLS treatment
* Placebo responders identified during the placebo run-in

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 731 (Actual)
Dates: Start 2008-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (88):
- United States (38):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Jasper, Alabama
  - Pfizer Investigational Site, Tuscaloosa, Alabama
  - Pfizer Investigational Site, Glendale, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Northridge, California
  - Pfizer Investigational Site, Redondo Beach, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Boca Raton, Florida
  - Pfizer Investigational Site, Hallandale, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Chevy Chase, Maryland
  - Pfizer Investigational Site, Newton, Massachusetts
  - Pfizer Investigational Site, Southfield, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Princeton, New Jersey
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Salisbury, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Lafayette Hill, Pennsylvania
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, Walla Walla, Washington
- Austria (3):
  - Pfizer Investigational Site, Innsbruck
  - Pfizer Investigational Site, Linz
  - Pfizer Investigational Site, Vienna
- Finland (4):
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Kuopio
  - Pfizer Investigational Site, Tampere
  - Pfizer Investigational Site, Turku
- Germany (26):
  - Pfizer Investigational Site, Achim
  - Pfizer Investigational Site, Bad Saarow
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bochum
  - Pfizer Investigational Site, Bremen
  - Pfizer Investigational Site, Dortmund
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Freiburg im Breisgau
  - Pfizer Investigational Site, Gelsenkirchen
  - Pfizer Investigational Site, Halle
  - Pfizer Investigational Site, Hamm
  - Pfizer Investigational Site, Jena
  - Pfizer Investigational Site, Jülich
  - Pfizer Investigational Site, Kassel
  - Pfizer Investigational Site, Köthen
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Marburg
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Oldenburg
  - Pfizer Investigational Site, Prien am Chiemsee
  - Pfizer Investigational Site, Schwerin
  - Pfizer Investigational Site, Siegen
  - Pfizer Investigational Site, Ulm
  - Pfizer Investigational Site, Unterhaching
  - Pfizer Investigational Site, Westerstede
  - Pfizer Investigational Site, Würzburg
- Italy (5):
  - Pfizer Investigational Site, Pavia
  - Pfizer Investigational Site, Pisa
  - Pfizer Investigational Site, Rome
  - Pfizer Investigational Site, Troina
  - Pfizer Investigational Site, Troina(EN)
- Netherlands (2):
  - Pfizer Investigational Site, Ede
  - Pfizer Investigational Site, Zwolle
- Spain (4):
  - Pfizer Investigational Site, Barcelona, Cataluña/Spain
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Granada
  - Pfizer Investigational Site, Madrid
- Sweden (5):
  - Pfizer Investigational Site, Avesta
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Örebro
  - Pfizer Investigational Site, Skövde
  - Pfizer Investigational Site, Stockholm
- Pfizer Investigational Site, Reading Berks, United Kingdom

REFERENCES:
- [Derived] Allen RP, Chen C, Garcia-Borreguero D, Polo O, DuBrava S, Miceli J, Knapp L, Winkelman JW. Comparison of pregabalin with pramipexole for restless legs syndrome. N Engl J Med. 2014 Feb 13;370(7):621-31. doi: 10.1056/NEJMoa1303646. PMID 24521108
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081186&StudyName=Long%20Term%20Study%20Of%20Pregabalin%20In%20Idiopathic%20Restless%20Legs%20Syndrome%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin 300 mg: Pregabalin (PGB) capsule 300 milligram (mg) once daily following a two week up escalation (Day 1-5: 75 mg once daily; Day 6-10: 150 mg once daily and Day 11 onwards: 300 mg once daily) up to 52 weeks along with placebo (PBO) capsule matched to PGB 300 mg in week 13 and 14. Participants were administered a tapering dose of PGB 150 mg once daily (Day 1-3); 75 mg once daily (Day 4-6) and matching PBO capsule once daily on Day 7 after completion of 52 weeks treatment.
- Pramipexole 0.25 mg: Pramipexole (PPX) 0.25 mg capsules administered once daily following a two week up escalation (Day 1-5: 0.125 mg once daily; Day 6 onwards: 0.25 mg once daily) up to 52 weeks along with PBO capsule matched to PPX 0.25 mg in week 13 and 14. Participants were administered a tapering dose of PPX 0.125 mg once daily (Day 1-3) and matching PBO capsule once daily (Day 4-7) after completion of 52 weeks treatment.
- Pramipexole 0.5 mg: PPX capsule 0.5 mg once daily following a two week up escalation (Day 1-5: 0.125 mg once daily; Day 6-10: 0.25 mg once daily and Day 11 onwards: 0.5 mg once daily) up to 52 weeks along with PBO capsule matched to PPX 0.5 mg in week 13 and 14. Participants were administered a tapering dose of PPX 0.25 mg once daily (Day 1-3); 0.125 mg once daily (Day 4-6) and matching PBO capsule once daily on Day 7 after completion of 52 weeks treatment.
- Placebo to Pregabalin 300 mg: PBO capsules matched to PGB 300 mg once daily following a two week up escalation (Day 1-5: 75 mg once daily; Day 6-10: 150 mg once daily and Day 11 onwards: 300 mg once daily) for 12 weeks, re-randomized to PGB 300 mg following a two week up escalation (Day 1-5: 75 mg once daily; Day 6-10: 150 mg once daily and Day 11 onwards: 300 mg once daily) up to 40 weeks. Participants were administered a tapering dose of PGB 150 mg once daily (Day 1-3); 75 mg once daily (Day 4-6) and matching PBO capsule once daily on Day 7 after completion of 52 weeks treatment.
- Placebo to Pramipexole 0.25 mg: PBO capsules matched to PPX 0.25 mg once daily following a two week up escalation (Day 1-5: 0.125 mg once daily and Day 6 onwards: 0.25 mg once daily) for 12 weeks, re-randomized to PPX 0.25 mg following a two week up escalation (Day 1-5: 0.125 mg once daily and Day 6 onwards: 0.25 mg once daily) up to 40 weeks. Participants were administered a tapering dose of PPX 0.125 mg once daily (Day 1-3) and matching PBO capsule once daily (Day 4-7) after completion of 52 weeks treatment.
- Placebo to Pramipexole 0.5 mg: PBO capsules matched to PPX 0.5 mg once daily following a two week up escalation (Day 1-5: 0.125 mg once daily; Day 6-10: 0.25 mg once daily and Day 11 onwards: 0.5 mg once daily) for 12 weeks, re-randomized to PPX 0.5 mg following a two week up escalation (Day 1-5: 0.125 mg once daily; Day 6-10: 0.25 mg once daily and Day 11 onwards: 0.5 mg once daily) up to 40 weeks. Participants were administered a tapering dose of PPX 0.25 mg once daily (Day 1-3); 0.125 mg once daily (Day 4-6) and matching PBO capsule once daily on Day 7 after completion of 52 weeks treatment.
Period: Overall Study
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo to Pregabalin 300 mg | Placebo to Pramipexole 0.25 mg | Placebo to Pramipexole 0.5 mg
Started | 185 | 183 | 182 | 61 | 59 | 61
Treated | 182 | 178 | 180 | 59 | 59 | 61
Completed | 93 | 82 | 89 | 32 | 29 | 29
Not Completed | 92 | 101 | 93 | 29 | 30 | 32
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Did not meet entrance criteria | 4 | 1 | 2 | 1 | 0 | 0
Not completed — Lack of Efficacy | 5 | 18 | 13 | 4 | 8 | 7
Not completed — Lost to Follow-up | 8 | 15 | 8 | 2 | 6 | 6
Not completed — Withdrawal by Subject | 14 | 17 | 9 | 2 | 5 | 3
Not completed — Other | 3 | 6 | 8 | 2 | 0 | 4
Not completed — Protocol Violation | 6 | 9 | 9 | 0 | 2 | 3
Not completed — Adverse Event | 52 | 35 | 44 | 17 | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo to Pregabalin 300 mg | Placebo to Pramipexole 0.25 mg | Placebo to Pramipexole 0.5 mg | Total
Number analyzed (Participants) | 182 | 178 | 180 | 59 | 59 | 61 | 719
Age, Customized [Number; unit: Participants]
  Less than 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18 to 44 years | 37 | 34 | 45 | 11 | 17 | 20 | 164
  45 to 64 years | 101 | 85 | 84 | 29 | 32 | 31 | 362
  Greater than and equal to 65 years | 44 | 59 | 51 | 19 | 10 | 10 | 193
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 108 | 99 | 37 | 36 | 38 | 441
  Male | 59 | 70 | 81 | 22 | 23 | 23 | 278

OUTCOME MEASURES:

1. Primary Outcome: Restless Legs Syndrome (RLS) Symptom Severity
Description: International Restless Legs Syndrome Study Group Rating Scale (IRLS) is psychometrically and clinically valid and reliable clinician-administered instrument used to assess the severity of RLS. It assesses RLS symptom severity and impact on daily living and is comprised of 10 items, scored on 0 to 4 scale, where lower score indicates lower symptom severity/impact on living. Two subscale scores are symptom severity (6 items) ranging from 0-24 (lower score indicates lower symptom severity) and impact on daily living (3 items) ranging from 0-12 (lower score indicates lower impact on living). Item 3 is unrelated to the other items. The global score is calculated from all 10 items, range from 0 to 40, where lower scores reflect lower severity and better quality of life.
Time Frame: Baseline
Population: Intent-to-treat (ITT) population included all randomized participants who took at least 1 dose of study medication and had at least one post-randomization efficacy assessment on any efficacy scale. Here, the 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure for each group respectively.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Placebo: PBO capsules matched to PGB 300 mg/ PPX 0.5 mg/ PPX 0.25 mg once daily following a two week up escalation for 12 weeks, re-randomized to 1 of the 3 active treatments (PGB 300 mg/ PPX 0.5 mg/ PPX 0.25 mg) and dose was escalated to the assigned fixed dose over 2 weeks and continued up to 40 weeks followed by dose tapering over 1 week similar to the active treatment.
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 177 | 169 | 178 | 172
Units on a Scale | 22.30 (5.73) | 22.40 (5.37) | 22.10 (5.19) | 22.40 (5.58)

2. Primary Outcome: Change From Baseline in the RLS Symptom Severity at Week 12
Description: IRLS is psychometrically and clinically valid and reliable clinician-administered instrument used to assess the severity of RLS. It assesses RLS symptom severity and impact on daily living and is comprised of 10 items, scored on 0 to 4 scale, where lower score indicates lower symptom severity/impact on living. Two subscale scores are symptom severity (6 items) ranging from 0-24 (lower score indicates lower symptom severity) and impact on daily living (3 items) ranging from 0-12 (lower score indicates lower impact on living). Item 3 is unrelated to the other items. The global score is calculated from all 10 items, range from 0 to 40, where lower scores reflect lower severity and better quality of life.
Time Frame: Baseline, Week 12
Population: ITT population included all randomized participants who took at least 1 dose of study medication and had at least one post-randomization efficacy assessment on any efficacy scale. Here, the 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure for each group respectively.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 177 | 169 | 178 | 172
Units on a Scale | -11.80 (0.47) | -7.90 (0.49) | -10.50 (0.47) | -7.30 (0.48)
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; For pregabalin 300 mg versus placebo: Mixed model analysis was used to analyze RLS symptom severity score with baseline value, region [United states (US) or European union (EU)], treatment, week and treatment by week interaction as fixed effects; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — This analysis was step 1 in a step-down procedure (if p<0.05, then continue to next step) used to control the Type I error rate. This procedure was stopped at Step 6. The analysis was done at a significance level of alpha = 0.05, 2-sided; Spatial power covariance structure was used; Least squares (LS) mean difference = -4.50, 95% CI 2-sided [-5.90 to -3.20], Standard Error of Mean 0.67
Statistical Analysis 2: Comparison: Pramipexole 0.25 mg vs Placebo; For pramipexole 0.25 mg versus placebo: Mixed model analysis was used to analyze RLS symptom severity score with baseline value, region (US or EU), treatment, week and treatment by week interaction as fixed effects; Test type: Superiority or Other; p = 0.3603, Mixed Models Analysis — This analysis was not included in the step-down procedure (if p<0.05, then continue to next step) to control Type I error. The analysis was done at a significance level of alpha = 0.05, 2-sided; Spatial power covariance structure was used; LS mean difference = -0.6, 95% CI 2-sided [-2.0 to 0.7], Standard Error of Mean 0.68
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; For pramipexole 0.5 mg versus placebo: Mixed model analysis was used to analyze RLS symptom severity score with baseline value, region (US or EU), treatment, week and treatment by week interaction as fixed effects; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; Spatial power covariance structure was used; LS mean difference = -3.2, 95% CI 2-sided [-4.5 to -1.9], Standard Error of Mean 0.67

3. Primary Outcome: Percentage of Participants Responding to Treatment at Week 12
Description: CGI-I: 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected. Responders were defined as participants who report CGI-I score of "very much improved" or "much improved".
Time Frame: Week 12
Population: ITT population. Last observation carried forward (LOCF) method was used. Here, 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure for each group respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 175 | 168 | 177 | 173
Percentage of participants | 71.40 | 51.20 | 62.70 | 46.80
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; For pregabalin 300 mg versus placebo: Cochran-Mantel-Haenszel (CMH) test stratified by geographical region (US or EU) was used to analyze CGI-I responder status; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — This analysis was step 2 in a step-down procedure (if p<0.05, then continue to next step) used to control the Type I error rate. This procedure was stopped at Step 6. The analysis was done at a significance level of alpha = 0.05, 2-sided
Statistical Analysis 2: Comparison: Pramipexole 0.25 mg vs Placebo; For pramipexole 0.25 mg versus placebo: CMH test stratified by geographical region (US or EU) was used to analyze CGI-I responder status; Test type: Superiority or Other; p = 0.4393, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; For pramipexole 0.5 mg versus placebo: CMH test stratified by geographical region (US or EU) was used to analyze CGI-I responder status; Test type: Superiority or Other; p = 0.0022, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 2]

4. Primary Outcome: Percentage of Participants With Augmentation
Description: Augmentation was worsening of RLS symptoms, attributable to a specific long-term therapeutic intervention for RLS. Percentage of participants with augmentation was evaluated by centralized evaluation board using a set of assessment criteria for potential augmentation which included structured interview for diagnosis of augmentation during RLS treatment (SIDA-RLS), augmentation severity rating scale (ASRS), clinical judgment. ASRS measures severity of augmentation and consist of three items to be completed by clinician. Clinician would score participants' answers by comparing post-baseline evaluations to those at baseline. ASRS total score range: 0-24, with higher score indicating more severe augmentation.
Time Frame: Baseline up to Week 52
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg
Number analyzed (Participants) | 176 | 167 | 178
Percentage of participants | 1.70 | 6.60 | 9.00
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Pramipexole 0.25 mg; For pramipexole 0.25 mg versus pregabalin 300 mg: Stratified log rank test by block (40 weeks versus 52 weeks of active treatment) was used to calculate p-value; Test type: Superiority or Other; p = 0.0826, Log Rank — This analysis was step 6 in a step-down procedure (if p<0.05, then continue to next step) used to control the Type I error rate. This procedure was stopped at Step 6. The analysis was done at a significance level of alpha = 0.05, 2-sided
Statistical Analysis 2: Comparison: Pregabalin 300 mg vs Pramipexole 0.5 mg; For pramipexole 0.5 mg versus pregabalin 300 mg: Stratified log rank test by block (40 weeks versus 52 weeks of active treatment) was used to calculate p-value; Test type: Superiority or Other; p = 0.0012, Log Rank — This analysis was step 3 in a step-down procedure (if p<0.05, then continue to next step) used to control the Type I error rate. This procedure was stopped at Step 6. The analysis was done at a significance level of alpha = 0.05, 2-sided

5. Secondary Outcome: Subjective Sleep Questionnaire (SSQ): Subjective Waking After Sleep Onset (WASO)
Description: SSQ: Participant-rated instrument used to assess previous night's sleep profile. It is used to measure sleep quantity and quality and is comprised of 5 items yielding 5 subscale scores: latency (1 item), hours of sleep (1 item), number of awakenings (1 item), total WASO (1 item), quality of sleep (1 item). WASO is time spent awake from sleep onset to final awakening. Total WASO subscale (in minutes): numerical rating completed by the participant 30 minutes after waking; recall period is the night before. Total WASO subscale score ranges from 0-1440 minutes. Lower value indicates better sleep.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 168 | 158 | 169 | 163
minutes | 90.60 (76.10) | 100.20 (85.92) | 83.90 (77.35) | 79.50 (69.85)

6. Secondary Outcome: Change From Baseline in SSQ: Subjective WASO at Week 12
Description: as for outcome 5
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 168 | 158 | 169 | 163
minutes | -49.86 (3.06) | -33.69 (3.15) | -37.18 (3.04) | -32.61 (3.10)
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; For pregabalin 300 mg versus placebo: Mixed model analysis was used to analyze SSQ-Subjective WASO score with baseline value, region (US or EU), treatment, week and treatment by week interaction as fixed effects; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — This analysis was step 7 in a step-down procedure (if p<0.05, then continue to next step) used to control the Type I error rate. This procedure was stopped at Step 6. The analysis was done at a significance level of alpha = 0.05, 2-sided; Spatial power covariance structure was used; LS mean difference = -17.25, 95% CI 2-sided [-25.76 to -8.74], Standard Error of Mean 4.332
Statistical Analysis 2: Comparison: Pramipexole 0.25 mg vs Placebo; For pramipexole 0.25 mg versus placebo: Mixed model analysis was used to analyze SSQ-Subjective WASO score with baseline value, region (US or EU), treatment, week and treatment by week interaction as fixed effects; Test type: Superiority or Other; p = 0.8075, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; Spatial power covariance structure was used; LS mean difference = -1.07, 95% CI 2-sided [-9.73 to 7.58], Standard Error of Mean 4.408
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; For pramipexole 0.5 mg versus placebo: Mixed model analysis was used to analyze SSQ-Subjective WASO score with baseline value, region (US or EU), treatment, week and treatment by week interaction as fixed effects; Test type: Superiority or Other; p = 0.2906, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; Spatial power covariance structure was used; LS mean difference = -4.57, 95% CI 2-sided [-13.05 to 3.91], Standard Error of Mean 4.318

7. Secondary Outcome: Subjective Sleep Questionnaire (SSQ): Latency Subscale Score at Week 12
Description: SSQ: Participant-rated instrument used to assess previous night's sleep profile. It is used to measure sleep quantity and quality and is comprised of 5 items yielding 5 subscale scores: latency (1 item), hours of sleep (1 item), number of awakenings (1 item), total WASO (1 item), quality of sleep (1 item). Latency subscale (in minutes): numerical rating completed by the participant 30 minutes after waking; recall period is the night before. Latency subscale score ranges from 0-840 minutes. Lower value indicates better sleep.
Time Frame: Week 12
Population: ITT population included all randomized participants who took at least 1 dose of study medication and had at least one post-randomization efficacy assessment on any efficacy scale. Here, 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure for each group respectively.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 169 | 161 | 174 | 165
minutes | 41.60 (35.76) | 43.10 (35.84) | 35.90 (33.08) | 47.70 (44.89)

8. Secondary Outcome: Subjective Sleep Questionnaire (SSQ): Hours of Sleep Subscale Score at Week 12
Description: SSQ: Participant-rated instrument used to assess previous night's sleep profile. It is used to measure sleep quantity and quality and is comprised of 5 items yielding 5 subscale scores: latency (1 item), hours of sleep (1 item), number of awakenings (1 item), total WASO (1 item), quality of sleep (1 item). Hours of sleep subscale: numerical rating completed by the participant 30 minutes after waking; recall period is the night before. Hours of sleep subscale score ranges from 0-16 hours. Higher value indicates better sleep.
Time Frame: Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 170 | 161 | 174 | 165
hours | 7.00 (1.05) | 6.70 (1.19) | 6.80 (1.09) | 6.70 (1.16)

9. Secondary Outcome: Subjective Sleep Questionnaire (SSQ): Number of Awakenings Subscale Score at Week 12
Description: SSQ: Participant-rated instrument used to assess previous night's sleep profile. It is used to measure sleep quantity and quality and is comprised of 5 items yielding 5 subscale scores: latency (1 item), hours of sleep (1 item), number of awakenings (1 item), total WASO (1 item), quality of sleep (1 item). Number of awakenings subscale: numerical rating completed by the participant 30 minutes after waking; recall period is the night before. Number of awakenings subscale score ranges from 0-30. Lower value indicates better sleep.
Time Frame: Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: awakenings
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 170 | 161 | 174 | 165
awakenings | 1.10 (1.14) | 1.70 (1.22) | 1.50 (1.08) | 1.80 (2.14)

10. Secondary Outcome: Subjective Sleep Questionnaire (SSQ): Quality of Sleep Subscale Score at Week 12
Description: SSQ: Participant-rated instrument used to assess previous night's sleep profile. It is used to measure sleep quantity and quality and is comprised of 5 items yielding 5 subscale scores: latency (1 item), hours of sleep (1 item), number of awakenings (1 item), total WASO (1 item), quality of sleep (1 item). Quality of sleep subscale: numerical rating completed by the participant 30 minutes after waking; recall period is the night before. Quality of sleep subscale score ranges from 0-100. Higher score indicates better quality of sleep.
Time Frame: Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 170 | 161 | 174 | 165
Units on a scale | 66.50 (20.00) | 57.40 (19.83) | 60.20 (19.43) | 57.70 (20.27)

11. Secondary Outcome: RLS-Next Day Impact (RLS-NDI)
Description: The RLS-NDI is a participant-rated instrument designed to assess daytime performance as related to RLS and the participant's previous night's sleep. The instrument consists of 14 items that encompass 5 domains: tiredness; emotional functioning; social functioning; cognitive functioning; and activities of daily living. There is also 1 global item assessing overall well -being. Each item is scored on a 0-10 numeric rating scale. Total score is the sum of scores from question 1 to 14. The total score ranges from 0 to 140 where higher scores indicate a more severe impact.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 26 | 30 | 34 | 31
Units on a Scale | 49.30 (22.03) | 51.90 (18.62) | 58.40 (20.27) | 50.00 (22.64)

12. Secondary Outcome: Change From Baseline in RLS-NDI at Week 12
Description: as for outcome 11
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 26 | 30 | 34 | 31
Units on a Scale | -8.10 (2.88) | -4.30 (2.65) | -14.50 (2.50) | -6.60 (2.68)
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; For pregabalin 300 mg versus placebo: Mixed model analysis was used to analyze RLS-NDI with baseline value, region (US or EU), treatment, week and treatment by week interaction as fixed effects; Test type: Superiority or Other; p = 0.7073, Mixed Models Analysis — This analysis was step 8 in a step-down procedure (if p<0.05, then continue to next step) used to control the Type I error rate. This procedure was stopped at Step 6. The analysis was done at a significance level of alpha = 0.05, 2-sided; Spatial power covariance structure was used; LS mean difference = -1.50, 95% CI 2-sided [-9.30 to 6.30], Standard Error of Mean 3.93
Statistical Analysis 2: Comparison: Pramipexole 0.25 mg vs Placebo; For pramipexole 0.25 mg versus placebo: Mixed model analysis was used to analyze RLS-NDI with baseline value, region (US or EU), treatment, week and treatment by week interaction as fixed effects; Test type: Superiority or Other; p = 0.5299, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; Spatial power covariance structure was used; LS mean difference = 2.4, 95% CI 2-sided [-5.1 to 9.9], Standard Error of Mean 3.78
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; For pramipexole 0.5 mg versus placebo: Mixed model analysis was used to analyze RLS-NDI with baseline value, region (US or EU), treatment, week and treatment by week interaction as fixed effects; Test type: Superiority or Other; p = 0.0354, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; Spatial power covariance structure was used; LS mean difference = -7.9, 95% CI 2-sided [-15.2 to -0.5], Standard Error of Mean 3.69

13. Secondary Outcome: Limb Pain-Visual Analog Scale (Limb Pain-VAS)
Description: 100 millimeter (mm) line (Visual Analog Scale) marked by participant. Intensity of pain range (over past week): 0 mm = no pain to 100 mm = worst possible pain.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 163 | 155 | 167 | 158
mm | 4.20 (2.70) | 4.30 (2.58) | 4.00 (2.53) | 4.10 (2.52)

14. Secondary Outcome: Change From Baseline in Limb Pain-VAS at Week 12
Description: 100 mm line (VAS) marked by participant. Intensity of pain range (over past week): 0 mm = no pain to 100 mm = worst possible pain. Change = observation mean minus baseline mean.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 163 | 155 | 167 | 158
mm | -3.20 (0.20) | -2.64 (0.20) | -2.75 (0.21) | -2.20 (0.20)
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; For pregabalin 300 mg versus placebo: Mixed model analysis was used to analyze limb pain-VAS with baseline value, region (US or EU), treatment, week and treatment by week interaction as fixed effects; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis — This analysis was step 9 in a step-down procedure (if p<0.05, then continue to next step) used to control the Type I error rate. This procedure was stopped at Step 6. The analysis was done at a significance level of alpha = 0.05, 2-sided; Spatial power covariance structure was used; LS mean difference = -1.00, 95% CI 2-sided [-1.55 to -0.45], Standard Error of Mean 0.280
Statistical Analysis 2: Comparison: Pramipexole 0.25 mg vs Placebo; For pramipexole 0.25 mg versus placebo: Mixed model analysis was used to analyze limb pain-VAS with baseline value, region (US or EU), treatment, week and treatment by week interaction as fixed effects; Test type: Superiority or Other; p = 0.1242, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; Spatial power covariance structure was used; LS mean difference = -0.43, 95% CI 2-sided [-0.99 to 0.12], Standard Error of Mean 0.282
Statistical Analysis 3: Comparison: Pramipexole 0.5 mg vs Placebo; For pramipexole 0.5 mg versus placebo: Mixed model analysis was used to analyze limb pain-VAS with baseline value, region (US or EU), treatment, week and treatment by week interaction as fixed effects; Test type: Superiority or Other; p = 0.0553, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; Spatial power covariance structure was used; LS mean difference = -0.55, 95% CI 2-sided [-1.12 to 0.01], Standard Error of Mean 0.287

15. Secondary Outcome: Severity of Augmentation Symptoms at Week 12
Description: ASRS measures severity of augmentation and consist of three items to be completed by clinician. Clinician would score participants' answers by comparing post-baseline evaluations to those at baseline. ASRS total score range: 0-24, with higher score indicating more severe augmentation.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 176 | 167 | 177 | 170
Units on a Scale | 0.90 (1.60) | 1.60 (2.29) | 1.30 (1.87) | 1.40 (1.95)

16. Secondary Outcome: Clinical Global Impressions-Severity (CGI-S) at Week 12
Description: CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal-not ill at all) to 7 (among the most extremely ill participants). Higher score = more affected.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 176 | 169 | 178 | 173
Units on a Scale | 2.90 (1.18) | 3.50 (1.22) | 3.10 (1.17) | 3.70 (1.17)

17. Secondary Outcome: Medical Outcomes Study-Sleep Scale (MOS-SS) at Week 12
Description: MOS-SS: Participant rated instrument to assess sleep quantity, quality; comprised of 12 items yielding 7 subscale scores: sleep disturbance, snoring, awakening short of breath/headache, sleep adequacy, somnolence, sleep quantity, optimal sleep, 2 composite index scores: sleep problems Index I, II. Sleep adequacy data was reported at week 12 and not for first 12 weeks (average). Subscale scores range: 0-100; exception quantity of sleep (range 0-24 hours). With exception of sleep quantity and sleep adequacy, higher scores reflect poorer sleep outcomes.
Time Frame: Week 12
Population: ITT population included all randomized participants who took at least 1 dose of study medication and had at least one post-randomization efficacy assessment on any efficacy scale. Here, 'n' is signifying those participants who were evaluable for particular category for each group respectively.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 177 | 169 | 178 | 174
Units on a Scale
  Sleep disturbance (n = 175, 169, 178, 171) | 30.50 (21.84) | 39.30 (23.72) | 34.40 (20.89) | 38.60 (21.43)
  Snoring (n = 172, 169, 178, 170) | 29.00 (27.50) | 25.80 (28.46) | 25.80 (25.81) | 24.60 (24.57)
  Awakening short of breath (n = 175, 169, 178, 171) | 10.50 (15.78) | 12.30 (17.09) | 13.80 (18.22) | 9.60 (15.13)
  Sleep adequacy (n = 128, 120, 133, 125 ) | 61.30 (28.57) | 54.80 (29.45) | 55.20 (27.87) | 50.00 (28.74)
  Somnolence (n = 175, 169, 178, 171) | 23.90 (17.57) | 27.60 (18.61) | 25.50 (18.67) | 26.00 (18.77)
  Sleep quantity (n = 175, 169, 178, 171) | 6.80 (1.08) | 6.50 (1.25) | 6.60 (1.16) | 6.50 (1.26)
  Sleep problem index I (n = 175, 169, 178, 171) | 29.40 (17.26) | 35.30 (18.82) | 33.40 (16.73) | 35.00 (16.54)
  Sleep problem index II (n = 175, 169, 178, 171) | 30.70 (17.15) | 36.60 (18.90) | 34.10 (17.05) | 36.30 (16.81)

18. Secondary Outcome: Number of Participants With Medical Outcomes Study-Sleep Scale (MOS-SS)- Optimal Sleep at Week 12
Description: MOS-SS: Participant rated instrument to assess sleep quantity, quality; comprised of 12 items yielding 7 subscale scores: sleep disturbance, snoring, awakening short of breath/ headache, sleep adequacy, somnolence, sleep quantity, optimal sleep, 2 composite index scores: sleep problems Index I, II. Optimal sleep subscale scores range: 0-1; Optimal sleep = 1 if 'Average hours sleep' = 7 or 8, is 0 if 'Average hours sleep' is non-missing and less than 7, and is missing if 'Average hours sleep' is missing. Higher scores reflect better sleep outcomes.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 128 | 120 | 132 | 125
Participants | 84 | 64 | 77 | 68

19. Secondary Outcome: Profile of Mood State (POMS) at Week 12
Description: POMS are participant-rated instrument comprising 6 sub-scales (tension-anxiety, depression-dejection, anger-hostility, vigor-activity, fatigue-inertia, and confusion-bewilderment) and each subscale comprising 5 items, on 'How you feel right now?' (Scale: 0=not at all, 1=a little, 2=moderately, 3=quite a bit, 4=extremely). All items were rated in the same direction except for vigor-activity. A total score is obtained for each scale. The range of total score is 0 - 100, with higher score indicating more mood disturbance.
Time Frame: Week 12
Population: Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis due to lack of sufficient knowledge as how to analyze mood data inferentially in RLS population.
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

20. Secondary Outcome: Restless Legs Syndrome-Quality of Life Scale (RLS-QoL) at Week 12
Description: RLS QoL: Participant rated instrument used to assess the impact of RLS on quality of life and health status function (symptom severity, daily activity, social functioning, sleep, concentrating and decision making, traveling, sexual activity, and work) yielding a summary score ranging from 0-100. Higher scores reflect better quality of life.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 173 | 169 | 176 | 168
Units on Scale | 77.75 (10.92) | 73.33 (13.02) | 75.48 (12.69) | 73.23 (13.98)

21. Secondary Outcome: Medical Outcomes Study-Short Form 36 (SF-36) at Week 12
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being (physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health); 2 summary scores (physical and mental component); and self evaluated change in health status (summary of health status). The score for subscale scores and 2 summary score is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Summary of health status is a 5-point Likert scale ranging from "0=much worse now" to "4=much better now". Higher subscale and summary score reflect better health status.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 175 | 168 | 178 | 171
Units on a Scale
  Physical functioning | 83.70 (18.30) | 81.90 (19.56) | 82.40 (19.98) | 83.00 (19.22)
  Role physical | 81.20 (20.75) | 79.60 (19.37) | 79.10 (20.71) | 81.50 (19.70)
  Bodily pain | 73.30 (20.51) | 65.20 (20.14) | 69.00 (20.40) | 65.50 (20.03)
  General health | 73.60 (18.37) | 69.80 (18.33) | 70.50 (17.68) | 72.80 (19.47)
  Vitality | 62.40 (19.27) | 59.00 (19.69) | 59.80 (20.17) | 59.30 (20.51)
  Social functioning | 87.20 (18.01) | 84.50 (18.14) | 84.00 (18.75) | 86.80 (18.37)
  Role emotional | 85.10 (18.91) | 83.90 (17.77) | 84.60 (18.09) | 87.00 (18.25)
  Mental health | 77.40 (16.13) | 74.60 (16.80) | 76.10 (16.29) | 78.70 (15.23)
  Summary physical score | 78.00 (16.50) | 74.20 (15.92) | 75.30 (16.43) | 75.70 (16.03)
  Summary mental score | 78.00 (15.73) | 75.50 (15.60) | 76.10 (15.32) | 78.00 (15.76)
  Summary of health status | 3.10 (0.47) | 3.10 (0.49) | 3.20 (0.54) | 3.10 (0.53)

22. Secondary Outcome: Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI-SHP) at Week 12
Description: WPAI: 6 question participant rated questionnaire to determine degree to which SHP affected work productivity while at work and outside of work. Four scores are derived: percentage of absenteeism and presenteeism (reduced productivity while at work), overall work impairment score combining absenteeism and presenteeism, percentage of impairment in activities performed outside of work. Score range: 0 (not affected/no impairment) to 10 (completely affected/impaired). WPAI outcomes expressed as impairment percentages with higher numbers indicating greater impairment and less productivity.
Time Frame: Week 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Percentage of impairment
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo
Number analyzed (Participants) | 177 | 169 | 178 | 174
Percentage of impairment
  Overall work (n= 10, 7, 11, 10) | 6.00 (9.66) | 5.70 (11.34) | 9.10 (20.71) | 14.60 (23.39)
  Activity (n= 18, 22, 25, 20) | 12.20 (19.27) | 20.90 (24.28) | 22.80 (23.01) | 23.00 (24.52)
  Work time missed (n= 10, 7, 11, 10) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 1.50 (3.62)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin 300 mg | Pramipexole 0.25 mg | Pramipexole 0.5 mg | Placebo to Pregabalin 300 mg | Placebo to Pramipexole 0.25 mg | Placebo to Pramipexole 0.5 mg
Serious Adverse Events (participants affected / at risk) | 9/182 | 12/178 | 9/180 | 5/59 | 2/59 | 0/61
Other Adverse Events (participants affected / at risk) | 134/182 | 110/178 | 118/180 | 42/59 | 34/59 | 41/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 300 mg (N=182) | Pramipexole 0.25 mg (N=178) | Pramipexole 0.5 mg (N=180) | Placebo to Pregabalin 300 mg (N=59) | Placebo to Pramipexole 0.25 mg (N=59) | Placebo to Pramipexole 0.5 mg (N=61)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Amaurosis fugax (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 2 | 0 | 0 | 0 | 0
Device dislocation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0 | 0 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neurological symptom (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bladder dysplasia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bladder calculus removal (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0
Spinal deformity correction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 300 mg (N=182) | Pramipexole 0.25 mg (N=178) | Pramipexole 0.5 mg (N=180) | Placebo to Pregabalin 300 mg (N=59) | Placebo to Pramipexole 0.25 mg (N=59) | Placebo to Pramipexole 0.5 mg (N=61)
Vertigo (Ear and labyrinth disorders) | 13 | 2 | 5 | 3 | 0 | 0
Vision blurred (Eye disorders) | 3 | 4 | 1 | 3 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 9 | 5 | 4 | 1 | 3
Constipation (Gastrointestinal disorders) | 14 | 3 | 2 | 5 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 9 | 10 | 2 | 5 | 5
Dry mouth (Gastrointestinal disorders) | 9 | 4 | 14 | 2 | 1 | 2
Nausea (Gastrointestinal disorders) | 11 | 18 | 26 | 3 | 3 | 4
Vomiting (Gastrointestinal disorders) | 3 | 4 | 10 | 3 | 2 | 5
Fatigue (General disorders) | 23 | 19 | 22 | 7 | 5 | 8
Irritability (General disorders) | 5 | 9 | 2 | 2 | 1 | 1
Oedema peripheral (General disorders) | 12 | 4 | 6 | 1 | 2 | 1
Cystitis (Infections and infestations) | 3 | 4 | 0 | 1 | 1 | 4
Influenza (Infections and infestations) | 9 | 13 | 3 | 4 | 8 | 7
Nasopharyngitis (Infections and infestations) | 19 | 20 | 17 | 3 | 3 | 9
Sinusitis (Infections and infestations) | 6 | 3 | 4 | 4 | 4 | 0
Urinary tract infection (Infections and infestations) | 6 | 2 | 6 | 3 | 3 | 2
Weight increased (Investigations) | 16 | 12 | 12 | 2 | 7 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 9 | 8 | 1 | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 15 | 13 | 2 | 4 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 4 | 1 | 3 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 7 | 7 | 4 | 2 | 1
Balance disorder (Nervous system disorders) | 2 | 2 | 1 | 4 | 0 | 0
Dizziness (Nervous system disorders) | 39 | 15 | 17 | 10 | 6 | 3
Headache (Nervous system disorders) | 22 | 30 | 35 | 9 | 6 | 12
Paraesthesia (Nervous system disorders) | 5 | 4 | 3 | 3 | 1 | 0
Somnolence (Nervous system disorders) | 32 | 12 | 14 | 7 | 4 | 5
Depression (Psychiatric disorders) | 10 | 4 | 7 | 3 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 7 | 0 | 4 | 1
Hypertension (Vascular disorders) | 7 | 6 | 4 | 1 | 3 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 3 | 0 | 0

LIMITATIONS AND CAVEATS:
Names of Daytime Function-Participant Reported Outcome (DF-PRO) and Limb Pain-Numerical Rating Scale (Limb Pain-NRS) were updated to RLS-NDI and Limb Pain-VAS respectively to reflect measurement appropriately.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.